CLINICAL TRIAL: NCT02055274
Title: A Randomized, Double-blinded, Multiple Ascending Dose Study in Patients With Early-stage Parkinson's Disease to Evaluate the Pharmacokinetics and Safety of LY03003 Following Intramuscular Injections
Brief Title: Pharmacokinetics and Safety Study of LY03003 in Patients With Early-stage Parkinson's Disease
Acronym: 03003MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LY03003
Record Dates: First submitted 2014-01-31; First posted 2014-02-05 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinsons
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LY03003 (Experimental): 4 Stable doses of LY03003 14, 28, 42 and 56 mg
  Interventions: Drug: LY03003
- Neupro (Active Comparator): Neupro patch 2 mg/24 hours in the first week, and then be titrated to 4, 6 and 8 mg/24 hours at weekly intervals
  Interventions: Drug: Neupro
- Neupro PK (Active Comparator): Neupro patch 2 mg/24hr in the first week then titrated to 4 and 6mg/24hr
  Interventions: Drug: Neupro

INTERVENTIONS:
Drug: LY03003
  Arms: LY03003
Drug: Neupro
  Arms: Neupro; Neupro PK

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (PK) of LY03003 following multiple escalating intramuscular injections, as compared to Neupro patch and to evaluate the safety and tolerability and preliminary efficacy of multiple ascending dose (MAD) of LY03003 following intramuscular injections.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has Idiopathic Parkinson's Disease defined by the cardinal sign, Bradykinesia, plus the presence of at least 1 of the following: resting tremor, rigidity, or impairment of postural reflexes, and without any other known or suspected cause of Parkinsonism
2. Subject is Hoehn & Yahr stage ≤3
3. Subject is male or female aged ≥18 years at Screening
4. Subject has a Mini Mental State Examination (MMSE) score of ≥25
5. Subject has a Unified Parkinson's Disease Rating Scale (UPDRS) motor score (Part III) of ≥10 but ≤30 at Screening

Exclusion Criteria:

1. Subject has atypical Parkinson's syndrome(s) due to drugs (e.g., Metoclopramide, Flunarizine), metabolic neurogenetic disorders (e.g., Wilson's Disease), Encephalitis, Cerebrovascular Disease, or Degenerative Disease (e.g., progressive Supranuclear Palsy)
2. Subject has a history of Pallidotomy, Thalamotomy, deep brain stimulation, or fetal tissue transplant
3. Subject has dementia, active psychosis or hallucinations, or clinically significant depression
4. Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (CSSRS) at Screening
5. Subject has a history of symptomatic orthostatic hypotension with a decrease of ≥20 mmHg in systolic blood pressure (SBP) or ≥10 mmHg in diastolic blood pressure when changing from supine to standing position after having been at supine position for at least 5 minutes within 28 days prior to the Screening Visit, or SBP less than 105 mmHg at study entry, or reports clinical signs of clinically significant orthostatic hypotension within 28 days prior to the Screening Visit.
6. Subject is receiving therapy with a dopamine agonist (DA) either concurrently or has done so within 28 days prior to the Screening
7. Subject is receiving therapy with 1 of the following drugs either concurrently or within 28 days prior to screening: MAO-B inhibitors, DA releasing agents, DA modulating agent, DA antagonists, neuroleptics, or other medications that may interact with DA function.
8. Subject is currently receiving central nervous system active therapy (e.g., sedatives, hypnotics, antidepressants, anxiolytics), unless the dose has been stable for at least 28 days prior to Screening Visit and is likely to remain stable for the duration of the study. Patients should not take those medications within 8 hours prior to clinical visits
9. Subject has a current diagnosis of epilepsy, has a history of seizures as an adult, has a history of stroke, or has had a transient ischemic attack within 1 year prior to Screening
10. Subject has a history of known intolerance/hypersensitivity to non-dopaminergic antiemetics, such as domperidone, ondansetron, tropisetron, and glycopyrrolate
11. Subject has any other clinically relevant hepatic, renal and cardiac dysfunction, or other medical condition or laboratory abnormality including abnormal plasma magnesium level, which would in the judgment of the investigator, interfere with the subject's ability to participate in the study
12. Subject has a history of significant skin hypersensitivity to adhesive or other transdermal preparations or recent unresolved contact Dermatitis (this item is specific for patients to be enrolled to part 2 of this study)
13. Subjects with C-reactive protein levels of 2x of upper limit of normal range
14. Female subjects who are pregnant or are breastfeeding or are of childbearing potential without adequate contraception.
15. Patients with a positive finding in drug screening test or alcohol test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Cmax for the Pharmacokinetics (PK) of LY03003 | 5 Weeks

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 5 Weeks
Preliminary efficacy evaluation will be carried out based on Unified Parkinson's Disease Rating Scale (UPDRS) motor score (Part III) | 5 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simon Li, Study Director — Luye Pharma Group Ltd.
Locations (5):
- United States (5):
  - Collaborative Neuroscience Network LLC, Long Beach, California
  - Compass Research LLC, Orlando, Florida
  - West Georgia Sleep Disorders Center and Neurology Associates, Douglasville, Georgia
  - Quest Research Institute, Bingham Farms, Michigan
  - PRA - CRI Lifetree, Marlton, New Jersey